CLINICAL TRIAL: NCT03216226
Title: A Phase 3, Randomized, Double-Blind, Parallel Group Safety Trial to Evaluate the Immunogenicity of Dasiglucagon and GlucaGen® Administered Subcutaneously in Patients With Type 1 Diabetes Mellitus (T1DM)
Brief Title: A Trial to Evaluate the Immunogenicity of Dasiglucagon and GlucaGen in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: SynteractHCR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-16136
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: Glucagon; Dasiglucagon
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — dasiglucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dasiglucagon (ZP4207) (Experimental): Repeated single fixed doses (s.c.injection) of dasiglucagon
  Interventions: Drug: dasiglucagon
- GlucaGen (Experimental): Repeated single fixed doses (s.c.injection) of GlucaGen
  Interventions: Drug: GlucaGen

INTERVENTIONS:
Drug: dasiglucagon — Glucagon Analog
  Other Names: ZP4207
  Arms: dasiglucagon (ZP4207)
Drug: GlucaGen — Native Glucagon
  Other Names: GlucaGen HypoKit
  Arms: GlucaGen

SUMMARY:
The trial's objective is to evaluate the immunogenicity of repeated single doses of dasiglucagon* and GlucaGen following subcutaneous (SC) administration in patients with type 1 diabetes mellitus (T1DM) and further to evaluate the safety and tolerability of dasiglucagon and GlucaGen.

*dasiglucagon is the proposed International Nonproprietary Name (pINN) for ZP4207

DETAILED DESCRIPTION:
Patients with T1DM were randomly assigned in a 1:1 ratio to receive 3 SC injections of either dasiglucagon (0.6 mg) or GlucaGen (1 mg), with 1 week between doses. Patients were followed for 15 weeks from the day of the first dose to assess the immune response. Patients with previous exogenic glucagon exposure were not excluded from the trial, but the information on previous glucagon administration was recorded to enable subgroup analyses. It was expected that 112 patients in total would be randomly assigned to treatment groups and treated. A total of 90 patients were expected to complete the trial (45 in each treatment arm). To qualify as completed, the patient had to be dosed according to the procedure described in the protocol and to have blood drawn for the antidrug antibody analyses as scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities (trial-related activities are any procedure that would not have been performed during normal management of the patient)
* Availability for the entire trial period
* Age between 18 and 70 years, both inclusive
* Male or female patients with T1DM for at least 1 year. Diagnostic criteria as defined by the American Diabetes Association
* Hemoglobin A1c (HbA1c) <10%
* Stable anti-diabetic treatment for at least 1 month (e.g. within 10% insulin dose adjustment)

Exclusion Criteria:

* Previous administration of dasiglucagon (previously referred to as ZP4207)
* Known or suspected allergy to trial medication(s) or related products
* History of anaphylaxis or symptoms of severe systemic allergy (such as angioedema)
* Previous participation (randomization) in this trial
* Females who are pregnant according to a positive pregnancy test, actively attempting to get pregnant, or are lactating
* Patients on a closed loop artificial pancreas
* Receipt of any investigational drug within 3 months prior to screening
* Active malignancy within the last 5 years
* Congestive heart failure, New York Heart Association class II-IV
* Inadequately treated blood pressure as defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥90 mmHg at screening
* Current bleeding disorder, including use of anticoagulant treatment
* Known presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma (i.e. insulin-secreting pancreas tumor)
* Known or suspected HIV infection
* Use of a systemic beta-blocker drug, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before Day 1 of this trial
* Use of systemic corticosteroids, anti-inflammatory biological agents, kinase inhibitors or other immune modulating agents within the last 3 months prior to screening
* Donation of blood or plasma in the past month, or in excess of 500 mL within 12 weeks prior to screening
* A positive result in the alcohol and/or urine drug screen at the screening visit. Significant history of alcoholism or drug abuse as judged by the investigator or consuming more than 24 g alcohol per day for men, or more than 12 g alcohol per day for women.
* Surgery or trauma with significant blood loss within the last 2 months prior to screening
* Use of prescription or non-prescription medications known to cause QT prolongation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Sylvest, MSc Pharm, Study Director — Zealand Pharma A/S
Locations (7):
- United States (2):
  - Compass Research, Orlando, Florida
  - Advanced Clinical Research, Meridian, Idaho
- CRC - Clinical Research Center, Medizinische Universität Graz, Graz, Austria
- Canada (3):
  - LMC Manna Research, Barrie
  - LMC Calgary, Calgary
  - LMC Diabetes & Manna Research, Toronto
- Diabeteszentrum Hamburg West, Gemeinschaftspraxis für Innere Medizin, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasiglucagon (ZP4207): 3 repeated doses (s.c.injection) of 0.6 mg dasiglucagon, with 1 week between each dose.
  dasiglucagon: Glucagon Analog
- GlucaGen: 3 repeated doses (s.c.injection) of 1.0 mg GlucaGen, with 1 week between each dose.
  GlucaGen: Native Glucagon
Period: Overall Study
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Started (Randomized) | 57 | 55
Randomized and Treated | 57 | 54
Completed | 52 | 50
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Patient unable to take time off work to come in for the third injection | 1 | 0
Not completed — Deviation from protocol window during visit as patient had to leave for work | 0 | 1
Not completed — Patient withdrawn prior to treatment. Patient veins unsuitable for blood draws | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the patients who were randomized and treated: 111 in total
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen | Total
Number analyzed (Participants) | 57 | 54 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 52 | 107
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.21) | 38.8 (13.65) | 42.1 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 41 | 32 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 50 | 52 | 102
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 28 | 26 | 54
  Austria | 15 | 15 | 30
  United States | 5 | 5 | 10
  Germany | 9 | 8 | 17
Body weight [Mean (Standard Deviation); unit: kg] | 82.9 (18.44) | 82.7 (16.25) | 82.8 (17.33)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (4.88) | 27.4 (4.70) | 27.3 (4.77)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With ADA
Description: Percentage of the combined results of treatment-induced ADA-positive patients and treatment-boosted ADA-positive patients out of the total number of evaluable patients. ADA = antidrug antibodies.
Time Frame: 104 days after the first dose
Population: Full analysis set of all patients in the safety analysis set (those randomized who received at least 1 dose of trial product) with at least 1 measurement of ADA titres at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 56 | 54
Participants
  Patients with ADA | 0 | 0
  Patients without ADA | 56 | 54

2. Secondary Outcome: Percentage of Patients With Treatment-induced ADA
Description: Percentage of the total number of evaluable patients that were ADA negative at baseline and ADA positive after drug administration out of the total number of evaluable patients. ADA = antidrug antibodies
Time Frame: 104 days after the first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 56 | 54
Participants
  Patients with ADA | 0 | 0
  Patients without ADA | 56 | 54

3. Secondary Outcome: Percentage of Patients With Treatment-boosted ADA
Description: Percentage of baseline ADA-positive patients with significant increases (≥5-fold) in ADA titre after drug administration out of the total number of evaluable patients. ADA = antidrug antibodies
Time Frame: 104 days after the first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 56 | 54
Participants
  Patients with ADA | 0 | 0
  Patients without ADA | 56 | 54

4. Secondary Outcome: Characterization of ADA Response - Neutralizing Activity
Description: Percentage of ADA positive patients with ADA neutralizing activity. ADA = antidrug antibodies.
Time Frame: 104 days after the first dose
Population: No ADAs were recorded in this trial, therefore it was not possible to characterize the ADA response.
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Characterization of ADA Response - Titer of Neutralizing Activity
Description: Titre of neutralizing activity of ADA positive patients. ADA = antidrug antibodies.
Time Frame: 104 days after the first dose
Population: No ADAs were recorded in this trial, therefore it was not possible to characterize the ADA response in terms of titre of neutralizing activity.
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Characterization of ADA Response - Cross-reactivity
Description: Percentage of ADA positive patients with cross-reactivity towards endogenous glucagon. ADA = antidrug antibodies.
Time Frame: 104 days after the first dose
Population: No ADAs were recorded in this trial, therefore it was not possible to characterize the ADA response in terms of cross-reactivity towards endogenous glucagon.
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Characterization of ADA Response - Timing
Description: The timing of detected ADA response. ADA = antidrug antibodies.
Time Frame: 104 days after the first dose
Population: No ADAs were recorded in this trial, therefore it was not possible to characterize the ADA response in terms of timing.
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Characterization of ADA Response - Duration
Description: The Duration of detected ADA response. ADA = antidrug antibodies.
Time Frame: 104 days after the first dose
Population: No ADAs were recorded in this trial, therefore it was not possible to characterize the ADA response in terms of duration.
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration Curve
Description: Area under the plasma concentration curve (AUC) 0-30 minutes at visit 2 and 4 (days 0 and 14). Plasma PK concentrations were measured before dosing and at 5, 10 and 30 minutes after dosing.
Time Frame: 0-30 minutes
Population: PK/PD set: all patients in the safety analysis set (patients who were randomized and received at least 1 dose of trial product) with at least 1 pre- and post-dose PK value at 1 visit. PK = pharmacokinetic. PD = pharmacodynamic.
Measure: Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
h*pmol/L
  Day 0 | 425 (220) | 548 (226)
  Day 14: number analyzed (Participants) | 52 | 49
  Day 14 | 499 (371) | 546 (181)

10. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration Curve
Description: Area under the plasma concentration curve (AUC) 0-90 minutes at visit 2 and 4 (days 0 and 14). Plasma PK concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 0-90 minutes
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
h*pmol/L
  Day 0 | 1560 (615) | 1290 (434)
  Day 14: number analyzed (Participants) | 52 | 49
  Day 14 | 1640 (611) | 1290 (379)

11. Secondary Outcome: Pharmacokinetics - Maximum Plasma Concentration
Description: Maximum plasma concentration (Cmax) at visit 2 and 4 (days 0 and 14). Plasma PK concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 90 minutes
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
pmol/L
  Day 0 | 1390 (609) | 1490 (537)
  Day 14: number analyzed (Participants) | 52 | 50
  Day 14 | 1820 (2460) | 1430 (498)

12. Secondary Outcome: Pharmacokinetics - Time to Maximum Plasma Concentration
Description: Time to maximum plasma concentration (Tmax) at visit 2 and 4 (days 0 and 14). Plasma PK concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 90 minutes
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
hours
  Day 0 | 0.5 [0.167 to 1.5] | 0.483 [0.0833 to 0.55]
  Day 14: number analyzed (Participants) | 52 | 50
  Day 14 | 0.5 [0.0833 to 1.5] | 0.5 [0.0833 to 0.517]

13. Secondary Outcome: Pharmacodynamics - Area Under the Effect Curve
Description: Plasma glucose profiles, area under the effect curve (AUE) 0-30 minutes at visit 2 and 4 (days 0 and 14). Plasma glucose concentrations were measured before dosing and at 5, 10 and 30 minutes after dosing.
Time Frame: 0-30 minutes
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
h*mmol/L
  Day 0 | 0.799 (0.449) | 0.886 (0.504)
  Day 14: number analyzed (Participants) | 52 | 48
  Day 14 | 0.869 (0.375) | 0.895 (0.511)

14. Secondary Outcome: Pharmacodynamics - Area Under the Effect Curve
Description: Plasma glucose profiles, area under the effect curve (AUE) 0-90 minutes at visit 2 and 4 (days 0 and 14). Plasma glucose concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 0-90 minutes
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
h*mmol/L
  Day 0 | 5.9 (2.42) | 5.86 (3.14)
  Day 14: number analyzed (Participants) | 52 | 49
  Day 14 | 6.47 (2.28) | 6.04 (2.63)

15. Secondary Outcome: Pharmacodynamics - Change From Baseline Plasma Glucose
Description: Change from baseline plasma glucose to maximum plasma glucose (CEmax) at visit 2 and 4 (days 0 and 14). Plasma glucose concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 90 minutes
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
mmol/L
  Day 0 | 6.25 (2.5) | 6 (3.01)
  Day 14: number analyzed (Participants) | 52 | 50
  Day 14 | 6.88 (2.43) | 6.21 (2.65)

16. Secondary Outcome: Pharmacodynamics - Time to Maximum Plasma Glucose Concentration
Description: Time to maximum plasma glucose concentration (Tmax) at visit 2 and 4 (days 0 and 14). Plasma glucose concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 90 minutes
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
hours
  Day 0 | 1.5 [0.0833 to 1.57] | 1.5 [0.483 to 1.6]
  Day 14: number analyzed (Participants) | 52 | 50
  Day 14 | 1.5 [0.167 to 1.58] | 1.5 [0.0833 to 1.52]

17. Secondary Outcome: Pharmacodynamics - An Increase in the Plasma Glucose Concentration of ≥20 mg/dL Within 30 Minutes After Treatment
Description: An increase in the plasma glucose concentration of ≥20 mg/dL within 30 minutes after treatment at visit 2 and visit 4. Plasma glucose concentrations were measured before dosing and at 5, 10, 30, 60 and 90 minutes after dosing.
Time Frame: 30 minutes
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
Number analyzed (Participants) | 57 | 54
Participants
  Day 0: Yes | 54 | 51
  Day 0: No | 3 | 3
  Day 14: number analyzed (Participants) | 52 | 49
  Day 14: Yes | 51 | 47
  Day 14: No | 1 | 2

ADVERSE EVENTS:
Time Frame: 104 days
Description: Adverse events were recorded at each trial visit by the investigator or other designated trial personnel.
Arm/Group | Dasiglucagon (ZP4207) | GlucaGen
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/54
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/54
Other Adverse Events (participants affected / at risk) | 42/57 | 43/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasiglucagon (ZP4207) (N=57) | GlucaGen (N=54)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasiglucagon (ZP4207) (N=57) | GlucaGen (N=54)
Hypoglycemia (Metabolism and nutrition disorders) | 27 (580) | 29 (447)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (8)
Nausea (Gastrointestinal disorders) | 26 (43) | 23 (33)
Vomiting (Gastrointestinal disorders) | 12 (18) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 6 (7) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 8 (14) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 2 (2) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Retinopathy (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT03216226/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03216226/SAP_003.pdf